CLINICAL TRIAL: NCT01894932
Title: Mindfulness-based Cognitive Group Therapy (MBCGT) and Psycho-physiological Stress Regulation Group for Depression and Psycho-physiological Stress Patient: An Outcome Study
Brief Title: MBCGT and Psycho-physiological Stress Regulation Group for Depression and Psycho-physiological Stress Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201103042RC
Record Dates: First submitted 2013-01-30; First posted 2013-07-10 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-07

CONDITIONS: Psychophysiologic Disorders; Stress, Psychological; Unipolar Depression
Keywords: Psychotherapy, Group
MeSH Terms: conditions — Psychophysiologic Disorders; Stress, Psychological; Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- MBCT Group for stress patient (Experimental): Mindfulness-based cognitive Group therapy will be administered on stress patient.
  Interventions: Behavioral: Mindfulness-based cognitive Group therapy
- MBCT Group for depression patient (Experimental): Mindfulness-based cognitive Group therapy will be administered on depression patient.
  Interventions: Behavioral: Mindfulness-based cognitive Group therapy
- SR group for stress patient (Experimental): psycho-physiological stress regulation group will be administered on stress patient.
  Interventions: Behavioral: psycho-physiological stress regulation group
- SR group for depression patient (Experimental): psycho-physiological stress regulation group will be administered on depression patients.
  Interventions: Behavioral: psycho-physiological stress regulation group
- normal (No Intervention): normal, no intervention.
- Drug treatment remission patient (No Intervention): Drug treatment remission patient

INTERVENTIONS:
Behavioral: Mindfulness-based cognitive Group therapy — In this study, groups of Mindfulness-based cognitive psychotherapy, will based on Segal, Williams & Teasdale (2002)'s work to redesigned an eight-week group course which adapted the local Taiwanese culture and add the appropriate revision of the content in a more easy to understand learning materials available to patient. The group would lead by 2 clinical psychologist and each session is about 2 hours.
  Arms: MBCT Group for depression patient; MBCT Group for stress patient
Behavioral: psycho-physiological stress regulation group — Physical and psychological stress regulation group in eight weeks, mainly to provide understanding of physical and mental effects of stress factors, self-conceptualization of stress and psychosomatic symptoms, physiological adjustment (relaxation, diet, exercise), psychological adjustment (positive primary, secondary assessment, cognitive identification), adjust negative thoughts, learn coping by using new choice. The group would lead by 2 clinical psychologist and each session is about 2 hours.
  Arms: SR group for depression patient; SR group for stress patient

SUMMARY:
Cases of physical and psychological stress problems is the need to prevent the risk of depression, primary care model will help to prevent depression. Many scholars have advocated for depression treatment not only concern symptom control and relief, prevention of recurrence should also be aware. The literature found cases had depression, with cognitive strategy bias , may cause recurrence of depression, under the influence of stress. The study was to assist the physical and mental disorder patient caused by stress and depression patient having cognitive and emotional regulation, and increased adapting Ability by ongoing two separate treatment groups ,Mindfulness-based Cognitive Group Therapy and psycho-physiological stress regulation Group Therapy. In addition, psychological groups can also help regulation daily Trivia stress, study will try to know about how group therapy's effects on patient's immune system.Research has three purposes,to validation 2 group model's results in assisting psycho-physiological stressed and depression patient, to establish group leader training center and prepare groups' standard procedure manuals,and to understand the patient's psycho-physical stress reaction on the immune system and fat cell hormone.

DETAILED DESCRIPTION:
The study was to assist the physical and mental disorder patient caused by stress and depression patient having cognitive and emotional regulation, and increased adapting Ability by ongoing two separate treatment groups ,Mindfulness-based Cognitive Group Therapy and psycho-physiological stress regulation Group Therapy. In addition, psychological groups can also help regulation daily Trivia stress, study will try to know about how group therapy's effects on patient's immune system.Research has three purposes,to validation 2 group model's results in assisting psycho-physiological stressed and depression patient, to establish group leader training center and prepare groups' standard procedure manuals,and to understand the patient's psycho-physical stress reaction on the immune system and fat cell hormone.

ELIGIBILITY:
Inclusion Criteria:

* Physical and mental condition caused by stress, physician diagnosed
* suffered from major depression, in remission more than three months , and had moderate or mild depressed mood

Exclusion Criteria:

* Suffering from schizophrenia or anxiety disorder .
* Chronic diseases (such as diabetes, stroke, heart disease, cancer, etc.) or major injury (such as a car accident brain injury)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-04; Primary Completion 2016-07 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
scores change on the Beck Depression Inventory, physical and psychological symptom score, negative self-thinking scale, mental focus and self-monitoring Scale, and Awareness Scale. | 25 weeks
  Self-administered questionnaire were seven parts, including: Beck Depression Inventory, physical and psychological symptom score, negative self-thinking scale, mental focus and self-monitoring Scale, Awareness Scale

CONTACTS AND LOCATIONS:
Overall Officials: Lue Bee-Horng, MD, Study Director — Department of Family Medicine, National Taiwan University Hospital
Locations (1):
- Department of Family Medicine, National Taiwan University Hospital, Taipei, Taiwan, Taiwan